CLINICAL TRIAL: NCT06773546
Title: Immunodysregulation As an Expression of Underlying Inborn Errors of Immunity: Implementation of Diagnostics and Management of Pediatric and Adult Patients with Immune System Disorders
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ID-TYPE
Record Dates: First submitted 2024-12-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Inborn Errors of Immunity
Keywords: Inborn errors of immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational, retro-prospective, moncentric study focused on Inborn Errors of Immunity, an heterogeneous group of inherited diseases due to defects in the differentiation and/or function of the immune system. The primary aim of this study is to obtain a clinical-immunological, functional and molecular characterisation of paediatric and adult patients with confirmed or suspected Inborn Errors of Immunity, particularly of patients with manifestations of immunedysregulation, focusing on clinical course, immunophenotypic laboratory and functional abnormalities, genetic background.

DETAILED DESCRIPTION:
Due to the observational nature of the study, patients were and will be treated according to normal clinical practice and in accordance with medical judgement. The following evaluations were performed in the retrospective cohort and will be performed in the prospective cohort:

* Standard haematochemical examinations;
* Extended lymphocyte typing;
* Plasma dosage of immunoglobulins;
* Evaluation of early and late responses to Measles-Parotitis-Rosolia and Diphtheria-Tetanus-Pertussis vaccinations;
* Evaluation of antibody responses to vaccines against Haemophilus Influenzae, Neisseria Meningitidis and Pneumococcus;
* Detection of auto-antibodies on HEp-2 cells, and of auto-antibodies directed against haemopoietic cells and proteins of innate and adaptive immunity;
* Plasma dosage of complement factors (C3, C4);
* Radiological assessment;
* Functional immunological assay;
* Molecular-genetic investigations of targeted gene panels involved in immunodysregulation and Inborn Errors of Immunity.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed or suspected Inborn Errors of Immunity;
* age < 50 years at onset of clinical features suspected for Inborn Errors of Immunity;
* obtaining informed consent from patients or parents/legal guardian of pediatric patients.

Exclusion Criteria:

• patients in whom infectious susceptibility and immunodysregulation can only be attributed to known non-immunological causes: acquired immunodeficiency secondary to chronic infections (HIV), and acquired immunodeficiency secondary to immunosuppressive treatment.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with confirmed or suspected Inborn Errors of Immunity, in particular patients with an immunodysregulated condition (autoimmunity, allergy, hyperinflammation and non-clonal lymphoproliferation, susceptibility to the development of malignant neoplasms) aged < 50 years at onset of clinical features suspected for Inborn Errors of Immunity, who referred to the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Category of diagnsoed Inborn Error of Immunity | at baseline
  categories I to X
Qualitative or quantitative alterations in innate immunity and/or adaptive immunity | at baseline
  presence or absence of alterations
Infective susceptibility | at baseline and every 6 months up to 1 year
  presence of one of the following conditions: invasive, severe, persistent, recurrent, opportunistic and/or vaccine strain infections
Immunodisregulation | at baseline and every 6 months up to 1 year
  presence of at least one disorder among atopy, hyperinflammation, autoimmunity, non-clonal lymphoproliferation and/or malignant neoplasms
Mortality | 1 year after diagnosis of Inborn Errors of Immunity
  time-to-event from diagnosis of Inborn Errors of Immunity up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Conti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bolgona, Italy